CLINICAL TRIAL: NCT05453318
Title: Efficacy and Acceptability of Thermal Ablation in the Treatment of Cervical Neoplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Referral Centre of Reproductive Health, Fez, Morocco (Unknown); Referral Centre of Reproductive Health, Taza, Morocco (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEC/09-22
Record Dates: First submitted 2022-06-22; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Cervical Neoplasm
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single arm study where women presenting with cervical lesions eligible to ablation were treated and followed-up for cure and adverse events.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thermal ablation Arm (Experimental): Treatment of cervical neoplasia by thermal ablation
  Interventions: Procedure: Treatment of cervical neoplasia by thermal ablation

INTERVENTIONS:
Procedure: Treatment of cervical neoplasia by thermal ablation — Women screened for cervical cancer by VIA presenting lesions eligible for ablative treatment were treated by thermal ablation. The treatment consisted in applying the probe on the lesion for 45 seconds at 100 degrees Celsius, with one to up to five applications depending on the lesion size. Following treatment, women were inquired about the pain level during the procedure, their satisfaction level of the procedure and whether they would recommend this treatment to their relatives. Women had a follow-up visit at 6 weeks to assess any complication of the procedure. Women were rescreened at 12 months, to evaluate the cure rate and any long-term adverse events.

SUMMARY:
Longitudinal study in two referral centers in Morocco to evaluate the effectiveness, the acceptability and safety of thermal ablation in the treatment of cervical neoplasia.

DETAILED DESCRIPTION:
The study population consisted of women with a positive Visual Inspection with Acetic Acid (VIA) screening test referred for ablative treatment. A total of 119 women with lesions eligible to ablative treatment were counselled and treated by thermal ablation. Informed consent was signed by each participant. Just after treatment, the patients were inquired about the level of pain during the procedure, and their level of satisfaction with the treatment. The women were followed-up at 6 weeks for any complication and re-assessed by colposcopy and biopsy at 12 months for any persistent or recurrent lesion and for any adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Women having been screened positive at VIA at the primary health center and referred to the diagnosis centre of Fez and Taza for ablative treatment by thermal ablation

Exclusion Criteria:

* Lesion occupying the 4 quadrants of the cervix
* Not visible squamous columnar junction (not Type 1 TZ (transformation zone))
* Vaginal or endocervical lesion
* Lesion subjective of cervical cancer

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Cure rate based on colposcopy and histology assessment | 1 year
  Cure rate is assessed after 1 year of treatment by colposcopy. Persistent or recurrent lesions are treated by thermal ablation, excision or hysterectomy according to the lesion size and characteristics.

SECONDARY OUTCOMES:
Acceptability of thermal ablation in terms of adverse events | 1 year
  Information on adverse events are collected immediately after the treatment, at the 6-week visit (short-term adverse events) and at the 12-month visit. Any minor and moderate complications are inquired.
Acceptability of thermal ablation in terms of satisfaction level | Within one hour after procedure
  Acceptability of thermal ablation is also measured by the satisfaction levelusing a nine-level Likert scale (from 1. Very unsatisfied to 9. Verysatisfied), through administration of a questionnaire just after treatment.
Safety of TA in terms of major adverse events | 1 year
  Information on adverse events are collected immediately after the treatment, at the 6-week visit (short-term adverse events) and at the 12-month visit. Any major complications (i.e. necessitating hospitalization) were inquired.

CONTACTS AND LOCATIONS:
Overall Officials: Zakia GHAFFOULI, MD, Principal Investigator — Diagnosis Centre, TAZA; Hanane BELCADI ABBASSI, MD, Principal Investigator — Diagnosis Centre, Fez
Locations (1):
- Referral Centre of Reproductive Health, Fes, Morocco

IPD SHARING:
Plan to Share IPD: No